CLINICAL TRIAL: NCT04066478
Title: Does Dehydroepiandrosterone (DHEA) Improve IVF Outcomes in Poor Responders? A Randomised, Double-blind, Placebo Controlled Trial
Brief Title: Does DHEA IVF Outcomes in Poor Responders?
Acronym: DHEA
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor
Sponsor: Homerton University Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017DHEA
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Infertility, Female; Poor Response to Ovulation Induction
MeSH Terms: conditions — Infertility, Female | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, placebo controlled study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teatment (Experimental): 75mg Dehydroepiandrosterone once daily for minimum ten weeks prior to starting ovarian stimulation
  Interventions: Drug: Dehydroepiandrosterone
- Comaprator (Placebo Comparator): 75mg placebo once daily for minimum ten weeks prior to starting ovarian stimulation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dehydroepiandrosterone — 75mg Dehydroepiandrosterone daily
  Arms: Teatment
Drug: Placebo — Placebo
  Arms: Comaprator

SUMMARY:
This study is a RCT to examine whether DHEA is capable of improving results for poor responders to ovarian stimulation during IVF treatment

DETAILED DESCRIPTION:
Poor responders to ovarian stimulation for IVF may be either predicted or evidenced from previous treatment. The ESHRE criteria for poor responders will be used to select candidates for this trial. A power calculation determined that 200 subjects should be recruited to each arm to receive either DHEA or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Markers for poor ovarian reserve (AMH <7 pmol/L(<1.1 ng/ml) and/or AFC< 7)
* Previous poor response to ovarian stimulation ( ≤3 oocytes with a conventional stimulation protocol)

Exclusion Criteria:

* Women > 42 years
* Women with premature ovarian failure / premature menopause (FSH>40 U/L). Women already taking DHEA.
* Patients with a known allergy to the trial drug or any of the active ingredients in the placebo.

Ages: 40 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-10-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rates | at 6-8 weeks gestation
  ultrasound confirmation of a foetus with a heartbeat

CONTACTS AND LOCATIONS:
Locations (1):
- Homerton Fertility Centre, London, United Kingdom